CLINICAL TRIAL: NCT06919081
Title: Phase II Study of the Efficacy of Topical Mesenchymal Stromal Cell Secretome for Ocular Surface Disease
Brief Title: Efficacy of Topical Mesenchymal Stromal Cell Secretome for Ocular Surface Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Eye Institute (NEI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ali R Djalilian, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1426; 3UH3EY031809-04S1 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Persistent Corneal Epithelial Defect; Corneal Epithelial Disorders
Keywords: persistent corneal epithelial disease/defects; persistent corneal epithelial; corneal epithelial disease; limbal stem cell deficiency; neurotrophic keratitis
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allogeneic Bone-Marrow Derived Mesenchymal Stromal Cells Secretome (Experimental): Allogeneic Bone-Marrow Derived Mesenchymal Stromal Cells Secretome for Topical Eye Drop
  Interventions: Drug: Allogeneic Bone-Marrow Derived Mesenchymal Stromal Cells Secretome
- Vehicle (Placebo Comparator): Vehicle (unconditioned media)
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Drug: Allogeneic Bone-Marrow Derived Mesenchymal Stromal Cells Secretome — Eye Drops
  Arms: Allogeneic Bone-Marrow Derived Mesenchymal Stromal Cells Secretome
Other: Vehicle Control — Eye Drops
  Arms: Vehicle

SUMMARY:
In this phase II randomized double-masked clinical trials, subjects with non-resolving corneal epithelial disease/defect (i.e., refractory to standard treatments for at least two weeks) will receive 8 weeks treatment of topical mesenchymal stem cell secretome or vehicle, with continued follow-up for up to Day 70.

ELIGIBILITY:
Inclusion Criteria:

* Age · Patients 18 years of age or older
* Ocular Health

  * Chronic corneal epithelial disease with fluorescein staining score 6 by NEI grading scale or persistent corneal epithelial defect present for longer than 14 days despite standard treatment
  * No objective clinical evidence of significant (> 50%) improvement/worsening of the epithelial disease in the last 14 days
  * Epithelial disease refractory to conventional non-surgical treatments (e.g., preservative-free artificial tears, gels or ointments; discontinuation of preserved topical drops; anti-inflammatory therapy)
  * If both eyes of subject meet the inclusion criteria, the eye with the higher fluorescein staining score will be enrolled to the study.
* Study Procedures

  * Only patients who satisfy all Informed Consent requirements may be included in the study. The patient and/or his/her legal representative must read, sign and date the Informed Consent document before any study-related procedures are performed. The Informed Consent form signed by patients and/or legal representative must have been approved by the UIC IRB for the current study. Patients must have the ability and willingness to comply with study procedures.

Exclusion Criteria:

* Ocular Health

  * Any active or suspected ocular infection (bacterial, viral, fungal or protozoal).
  * History of any ocular surgery (including laser or refractive surgical procedures) in the study eye within the 3 months prior to study enrollment.
  * Treatment with Oxervate in the study eye within 12 months of enrollment.
* Study Procedures

  * Known hypersensitivity to one of the components of the study or procedural medications (e.g., fluorescein).
  * Use of any investigational agent within 4 weeks of screening visit.
  * Participation in another clinical study at the same time as the present study.
  * Participants who are pregnant at the time of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Improvement of Corneal Epithelial Barrier and/or Integrity (Efficacy Outcome) | Baseline to Day 56
  Proportion of subjects with improved epithelial barrier and/or integrity from baseline to DAY 56 as determined by the investigator on slit lamp examination: · Improved epithelial barrier, defined as ³ 50 % improvement in corneal fluorescein staining score using NEI grading scale · Improved epithelial integrity, defined as complete closure of persistent epithelial defect, measured with ImageJ on slit lamp images

SECONDARY OUTCOMES:
Visual Acuity | Baseline to Day 56
  Percent change in best-corrected distance visual acuity from baseline to DAY 56 as measured using standard ETDRS protocols
Corneal staining and NEI grading | Baseline to Day 70
  Grading of fluorescein staining of the cornea Minimum score = 0 Maximum score = 15 Lower score is better
Ocular Surface Parameters | Baseline to Day 70
  Changes in ocular surface disease index (OSDI) from baseline to DAY 56 and DAY 70 Minimum value = 0 Maximum value = 100 Lower value is better
Corneal Epithelial Thickness | Baseline to Day 70
  Percent change in corneal epithelial thickness from baseline to DAY 56 and DAY 70, as measured by anterior segment OCT (AS-OCT)
Subject Symptoms | Baseline to Day 70
  Changes in ocular discomfort visual analog scale (VAS) 0 - 100, where 0 is no discomfort and 100 the worst discomfort, from baseline to DAY 70
Time to epithelial healing | Baseline to Day 70
  Time of improvement of epitheliopathy
Corneal Opacities/Scars | Baseline to Day 56
  Change in the size of corneal opacities and scars (if present) from baseline to DAY 56 as documented by slit lamp photographs
Corneal vascularization | Baseline to Day 56
  Change in corneal vascularization on slit lamp photographs from baseline to DAY 56
Conjunctival injection | Baseline to Day 56
  Change in conjunctival injection on slit lamp examination from baseline to DAY 56
Subbasal corneal nerve density | Baseline to Day 56
  Changes in subbasal corneal nerve density on confocal microscopy from baseline to Day 56
Ocular Surface Parameters | Baseline to Day 70
  Changes in Lissamine green staining from baseline to DAY 56 and DAY 70
Ocular Surface Parameters | Baseline to Day 70
  Changes in anesthetic Schirmer's test from baseline to DAY 56 and DAY 70

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Djalilian, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States